CLINICAL TRIAL: NCT02176434
Title: Pilot Feasibility Study of Combined Kidney and Hematopoietic Stem Cell Transplantation to Cure End-stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: swisstolerance.ch
Record Dates: First submitted 2014-06-23; First posted 2014-06-27 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; Transplantation; Tolerance
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolerance (Experimental): Combined kidney and hematopoietic stem cell transplantation from the same donor.
  Interventions: Procedure: Kidney and hematopoietic stem cell transplantation; Biological: hematopoietic stem cell

INTERVENTIONS:
Procedure: Kidney and hematopoietic stem cell transplantation — Kidney transplantation (day 0) Induction therapy (s. above) Hematopoietic stem cell transplantation (s. above)
Biological: hematopoietic stem cell

SUMMARY:
This pilot study of combined kidney and hematopoietic stem cell transplantation attempts to establish a protocol to induce immunological tolerance as a new strategy to prevent renal graft rejection. If successful, this strategy would restore renal function, while avoiding the risks associated with long-term standard anti-rejection therapy, and would represent the first option to cure end-stage renal disease.

DETAILED DESCRIPTION:
Trial design This is an open-label feasibility study of combined Human Leukocyte Antigen (HLA)-matched sibling hematopoietic stem cell and kidney transplantation. The study will be performed at the University Hospital of Zurich. The pilot study will include 5 to 8 donors and 5 to 8 recipients. We expect that 4 out of 5 recipients should be off immunosuppressive therapy at 6-12 months.

Study protocol

1. Non-study-specific interventions before transplantation Donor and recipients will be screened according to the established internal guidelines for living donor kidney and hematopoietic stem cell transplantation of the Transplantation Center of the University Hospital Zurich.
2. Study-specific interventions before transplantation

   * Potential candidates will be informed about this study by the treating physician. Interested patients will be informed in details about the study protocol, the potential benefits and risks. The patient will have sufficient time to decide to participate to this study or to undergo standard transplantation, to read and sing the informed consent form.
   * Total lymphoid irradiation: for the optimal planning of the total lymphoid irradiation, a mapping CT will be performed 2-4 weeks before therapy and repeated on day 1 after kidney transplantation.
   * Blood draw for establishment of chimerism determination.
   * The recipient will undergo one leukapheresis procedure before starting the conditioning regimen in order to bank cells for future scientific studies.
   * Stem cell mobilization and isolation in the donor by leukapheresis will be performed according to the standard protocols of the Stem cell transplantation center of the University Hospital Zurich
   * Donor-derived hematopoietic progenitor cells will be isolated from peripheral leukocytes by positive selection (CD34+ cells) using the Magnetic-Activated Cell Sorting (MACS) technology according to SOPs of the certified hematology laboratory of the University Children's Hospital Zurich. CD34 negative cells will be analyzed by Fluorescence-Activated Cell Sorting (FACS) to determine the amount of CD3 positive cells. Stem cells and flow through will be frozen until the transplant according to standard operating procedure (SOP) at the stem cell transplantation center at the University Hospital Zurich.
   * Since irradiation might reduce fertility the possibility of sperm conservation before transplantation will be offered to male recipients.
3. Induction protocol

   * Kidney transplantation (day 0)
   * A CT scan will be performed at day 1 after transplantation for a correct definitive plan of the irradiation protocol.
   * Immunosuppression: in the first weeks after kidney transplantation the recipients will be treated with standard immunosuppression, including methylprednisolone, prednisone, mycophenolate mofetil and cyclosporine A.
   * Additionally the patient will be treated with:

   Rabbit anti-thymocyte globulin (ATG): Thymoglobuline® 1.5 mg per kg; 5 daily injections from day 0 to day 4.

   Total lymphoid irradiation: 10 doses of 120 centigray (cGy) (total dose 12 Gy) each to the supradiaphragmatic lymph nodes, thymus, subdiaphragmatic lymph nodes and spleen; 10 daily doses from day 1 to day 11.

   • Hematopoietic stem cell transplantation (day 11 after kidney transplantation): Infusion of isolated CD34+ hematopoietic progenitor cells (≥10x10^6 cells/kg) Additionally the patients will receive 1x10^6 CD3+ T cells / kg body weight from the CD34- fraction to promote the engraftment of hematopoietic progenitor cells (T cell add-back)
4. Immunosuppression and anti-microbial prophylaxis

   * Methylprednisolone: steroids will be rapidly tapered during the first days after transplantation. All patients will be off of steroids at day 14.
   * Mycophenolate mofetil: 2 g per day, started at day 11 (4 to 6 hours after stem cell transplantation) and discontinued 1 month after stem cell transplantation.
   * Cyclosporine A:

First 3 months: whole blood through level (C0) 250-300 µg/ml

Month 3-6: cyclosporine will be tapered and discontinued at about 6 months if following criteria will be fulfilled:

* Sustained chimerism for at least 180 days
* No clinical signs of rejection
* Protocol biopsy showing no evidence of acute or chronic rejection
* No clinical signs of graft versus host disease
* Anti-microbial prophylaxis:

Amoxicillin/clavulanic acid 2.2 g preoperatively Sulfamethoxazole/Trimethoprim for 6 months Valganciclovir: a) low risk (D-R-) - no prophylaxis; b) intermediate risk (R+) - prophylaxis with valganciclovir 450mg once daily, starting after 1 month post transplant; c) high risk (D+R-) - prophylaxis with valganciclovir 450mg once daily, starting immediately after transplantation.

5 Post-operative monitoring

* Donor and recipient will be followed life-long in the outpatient clinic of the nephrology division according to local practice. During immunosuppression tapering and in the first months off of immunosuppression renal function will be closely monitored for an early detection of rejection episodes. Therefore, to participate to the study the patient has to agree with a weekly creatinine testing, which might also be performed by the patient's family doctor.
* Graft versus host disease will be monitored clinically at each regular visit as well as by measurement of liver function tests.
* The donor will be included in the control program of stem cells donors and living kidney donors as for regular transplant procedures (national registries for living kidney and stem cell donors)
* Chimerism level in peripheral blood will be regularly assessed
* Kidney allograft biopsies will be performed 6 months (before withdrawing of cyclosporine A) and 1 year after transplantation
* Immune reconstitution will be analyzed by FACS of peripheral blood leukocytes and additional functional assays in vitro.
* Functional immunological tolerance will be measured in in vitro assays after 1, 2, 6, 12, 18 and 24 months. These additional tests are of scientific interest, but will not influence clinical patient management.
* Quality of life will be assessed as routinely performed in the context of the Swiss transplant cohort study (www.stcs.ch)
* Regular monitoring for cancer development as done after conventional transplantation (skin cancer, breast cancer, prostate cancer).

Duration of subject participation and follow-up The active portion of this trial will begin approximately 2 months prior to the transplantation and continue until 2 years post-transplant. Study-related data will be collected for a minimum of 2 years post-transplant. All subjects will be followed indefinitely for graft and patient survival in routine clinical follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who are eligible for kidney transplantation
* Males or females 18 - 70 years of age.
* Subjects must have an HLA-matched sibling donor 25-70 years of age
* Men and women of reproductive potential must agree to use a reliable method of birth control
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Evidence of uncontrolled active infection (including replicating HIV, Hepatitic B and Hepatitis C) as defined by:

  1. clinical syndrome consistent with viral or bacterial infection, or
  2. fever with a clinical site of infection identified, or
  3. microbiologically documented infection
* Contraindication to therapy with any one of the proposed agents (e.g. allergy to ATG).
* Serologic positivity to HIV.
* Women of childbearing age in whom adequate contraception cannot be maintained, pregnant women or nursing mothers.
* Malignancy within the past two years, for which waiting time for transplantation is required by PENN registry consult, thereby excluding non-melanoma skin cancer and carcinoma in situ of the cervix.
* Liver transaminases > 3 x normal value.
* Cardiac ejection fraction < 50% by radionuclide ventriculography or echocardiography.
* Forced Expiratory Volume (FEV1) < 50% predicted or corrected Diffusing Capacity for Carbon Monoxide (DLCO) < 50 % predicted.
* Blood group incompatibility in the host-vs-graft direction.
* High risk of primary kidney disease recurrence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-09; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Renal allograft acceptance and ability to discontinue immunosuppressive therapy at 1 year | 1 year
  * Renal function as determined by eGFR (CKD-EPI) and proteinuria after discontinuation of immunosuppressive therapy (1 year after transplantation)
  * Evidence for rejection according to Banff classification, as assessed in the transplant biopsy performed after discontinuation of immunosuppressive therapy (1 year after transplantation)

SECONDARY OUTCOMES:
Engraftment of hematopoietic stem cells (chimerism) | 6 months
  Hematopoietic chimerism will be determined by measurement of donor-derived cells in peripheral blood
Absence of graft versus host disease | 6 and 12 months
  Presence and grade of graft versus host disease will be assessed by clinical evaluation
Absence of renal allograft rejection | 6 and 12 months
  Renal allograft rejection will be assessed by measurement of renal function (eGFR CKD-EPI) and proteinuria in kidney transplant biopsy performed at 6 months and 1 year after transplantation
T cell recovery and immune reconstitution | 6 and 12 months
  T cell recovery and immune reconstitution will be measured by FACS analysis of peripheral blood samples and by functional immunological tests in vitro (T cell proliferation, T cell toxicity)
Absence of opportunistic infections (immune competence) | 6 and 12 months
  Opportunistic infections will be monitored clinically as a surrogate of immune competence
Quality of life (questionnaire) | 6 and 12 months
  Quality of life will be assessed by a standardized validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ferh, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scandling JD, Busque S, Shizuru JA, Engleman EG, Strober S. Induced immune tolerance for kidney transplantation. N Engl J Med. 2011 Oct 6;365(14):1359-60. doi: 10.1056/NEJMc1107841. No abstract available. PMID 21991976